CLINICAL TRIAL: NCT04844489
Title: Study of the Humoral Response to SARS-CoV-2 Variants and of the Cellular Response After Vaccination Against COVID-19 in Immunocompromised People
Acronym: COVIVAC-ID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP210305; 2021-A00469-32 (Other: IDRCB)
Record Dates: First submitted 2021-04-02; First posted 2021-04-14 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2021-06

CONDITIONS: Autoimmune or Autoinflammatory Diseases; HIV; Multiple Sclerosis; Solid Tumors or Cancers; Solid Organ Transplant
Keywords: Covid-19; Vaccination; Variants; Neutralizing antibodies; Cellular immunity
MeSH Terms: conditions — Multiple Sclerosis; Neoplasms; COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood samples (Other)
  Interventions: Other: Blood samples for the study of the humoral response to SARS-CoV-2 variants and of the cellular response after vaccination against COVID-19

INTERVENTIONS:
Other: Blood samples for the study of the humoral response to SARS-CoV-2 variants and of the cellular response after vaccination against COVID-19 — Blood samples at:
  * D0 (the day of the injection of the SARS-CoV-2 vaccine),
  * during the 2nd injection as part of the national vaccination campaign (on D28)
  * during the 3rd injection for patients for whom a third injection is recommended (according to the recommendations in force)
  * then to M1, M6 and M12 of the last injection

SUMMARY:
Prospective, multicenter, non-comparative cohort study of immunocompromised people vaccinated against Covid-19 with the aim to know the humoral and cellular response to BNT162b2 vaccination against SARS-CoV-2 variants. This study will enroll patients in 5 parallel sub-cohorts of the same size, distinct according to the source of the immunosuppression: autoimmune or auto-inflammatory disease, HIV infection, multiple sclerosis, solid cancer, organ transplantation with prospective data collection and constitution of biological collections.

DETAILED DESCRIPTION:
The SARS-CoV-2 pandemic represents an extraordinary challenge for global health, it has caused more than 97 million cases of Covid-19 and 2 million deaths worldwide as of January 22, 2021. Vaccination against Covid-19 is an essential weapon to mitigate the consequences of the SARS-CoV-2 pandemic. Its effect in reducing mortality is of course expected in people most vulnerable to Covid-19 such as immunocompromised people.

In general, the immunogenicity of vaccines in immunocompromised populations is conditioned by the nature and intensity of the chronic pathology (s), the age and the treatments received. In addition, the emergence of new variants of SARS-CoV-2 is a major concern today. Three new variants that have rapidly become dominant within their countries have aroused concerns: B.1.1.7 (also known as VOC-202012/01), 501Y.V2 (B.1.351), and P.1 (B.1.1.28.1) and questions are raised about their potential to escape from vaccine-induced immunity. It is therefore important to be able to assess vaccine efficacy in subjects who are fragile with respect to these variants.

The investigators are proposing the establishment of a multicenter cohort study of immunocompromised people vaccinated against Covid-19 with the aim to know the humoral and cellular response to BNT162b2 vaccination against SARS-CoV-2 variants. The primary objective is to evaluate the neutralizing capacity of the antibodies regarding different variants of SARS-CoV-2 after vaccination on 1 month after the first injection, then on 1, 6 and 12 months after the last injection. In-depth immunophenotyping of immune blood cells which analyzes in detail the subpopulations of T lymphocytes and their responses to SARS-CoV-2 will be also analyze before vaccination and after vaccination on 1 month after the first injection, then on 1 month after the last injection. Extensive explorations of the humoral and cellular response to BNT162b2 vaccination will provide crucial data on the potential efficacy of the BNT162b2 vaccine on the recently identified SARS-CoV-2 variants, as well as innovative data on the dynamic of the functional responses of T cells and of the TCR repertoire, the dynamic of which (increase after vaccination, remote contraction) makes it possible to link them to a vaccine response, as has already been done in the context of other vaccination.

This study will provide a better understanding of the biological response to BNT162b2 vaccination in immunocompromised people with respect to the English VOC 202012/01, South African 501Y.V2 variants and any other variants that may emerge. In particular, the investigators are waiting to be able to estimate the proportion of patients whose immunogenicity suggests a reduction in the frequency of severe forms of COVID-19. Conversely, the investigators are waiting to estimate the proportion of patients with a level of immunogenicity too low to hope for good clinical protection against COVID-19. In addition, there are no data on the durability of the biological response to BNT162b2 vaccination.

It is possible that these observations could lead to the implementation of reinforced vaccination protocols for this population, as is already the case for vaccination for hepatitis B vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Patients eligible for BNT162b2 vaccination
* Immunocompromised patients according to one of the following criteria:

  1. Patients with autoimmune or autoinflammatory diseases treated

     1. For at least three months
     2. Having received at least 0.1 mg / kg / day of prednisone (or equivalent) for at least three months
     3. Currently receiving at least 5 mg / day of prednisone in combination with an immunosuppressant (methotrexate, cyclosporine, mycophenolate mofetil, rapamycin, azathioprine, cyclophosphamide) or biotherapy (anti-B cells (rituximab and others) anti-TNF, IL- 1, IL-6R, IL-12/23, IL-17, or B7 (CTLA4-Ig)) or a kinase inhibitor (Janus, Tyrosine))
  2. HIV-infected patients with a CD4 count <500 / mm3 and a viral load <50 copies / ml on stable antiretroviral therapy for at least 3 months
  3. Patients with multiple sclerosis treated with a disease-modifying drug for at least 3 months at a stable dose (teriflunomide, dimethyl-fumarate, fingolimod, ocrelizumab, rituximab, natalizumab)
  4. Patients with solid tumors or cancers:

     1. Patients who have received active cancer treatment other than chemotherapy (targeted therapy, radiotherapy, surgery, hormone therapy) in the previous month
     2. Patients who have received active cancer treatment with chemotherapy (alone or in combination with immunotherapy, radiotherapy or targeted therapy) in the previous month
     3. Patients who have received active oncology treatment with one or more immunotherapy (s) in combination with anti-PD1, anti-PD-L1, anti-CTLA4 antibodies without chemotherapy in the previous month.
  5. Solid organ transplant patients for more than 3 months who have not received a depleting T agent in the induction protocol, and for> 6 months otherwise
* Life expectancy of more than 3 months
* Having been informed about the study and having given their written and informed consent
* Beneficiaries or beneficiaries of a social security scheme

Exclusion Criteria:

* Patients who may be included in more than one of the sub-cohorts
* Other vaccination received in the 15 days preceding recruitment or planned in the month following the second vaccine injection
* Known or suspected allergy to one of the components of the vaccine
* Severe reaction after previous administration of any influenza vaccine (multiple sclerosis, Guillain-Barré syndrome)
* Contact subjects of a patient with an undetected documented SARS-CoV-2 infection
* Evocative signs of COVID-19
* History of documented SARS-CoV-2 infection of less than 3 months (RT-PCR, Lamp PCR, antigen test)
* Last outbreak of the disease less than 3 months old for patients with Multiple Sclerosis; less than a month old for patients with autoimmune or autoinflammatory diseases
* For patients with HIV, transient viremia (blip) less than 3 months old
* Intercurrent infection
* For organ transplants, episode of cellular or humoral rejection during the 3 months preceding inclusion
* Healthy volunteers
* Pregnancy less than 13 weeks old according to the declaration of pregnancy
* Refusal of participation by the patient
* Patients subject to legal protection measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a neutralizing antibody titer greater than 1/10 towards the wild strain and the English VOC 202012/01, South African 501Y.V2 variants and any other variants that may emerge | At the third injection visit and at one, six and twelve months after the last injection

SECONDARY OUTCOMES:
Proportion of patients with a positive serology by detection of IgG anti-receptor-binding domain (RBD) antibodies to the Spike protein of SARS-CoV-2 measured by the SARS-CoV technique -2 IgG II Quant assay (Abbott) | At second and third injection visits and at one, six and twelve months after the last injection
Proportion of patients with a positive serology by detection of the anti-Spike protein IgG antibodies of SARS-CoV-2 measured by the Euroimmun technique | At second and third injection visits and at one, six and twelve months after the last injection
Proportion of patients with positive anti-RBD IgG serology on D0 | At inclusion visit
Anti-RBD IgG level | At second and third injection visits and at one, six and twelve months after the last injection
Antibody neutralization title | At second and third injection visits and at one, six and twelve months after the last injection
Neutralization title for antibodies against the wild strain and to the English VOC 202012/01, South African 501Y.V2 variants and any other variants that could be introduced to emerge. | At second and third injection visits and at one, six and twelve months after the last injection
Supervised and unsupervised analyzes of deep immunophenotyping of T and B lymphocytes | At Day 0, at the third injection visit and at one month after the last injection
  Count of CD4 / CD8, B and NK T lymphocyte populations and quantification of Treg lymphocytes on fresh cells. In-depth immunophenotyping of T lymphocytes with naive distributions / memories and activation markers and on naive B distributions / memories and other classically described subpopulations
Cytometric measurement of intracellular cytokines (IFN, TNF, IL-2, IL4, IL10, IL-17) after stimulation of T lymphocytes by pools of SARS-CoV-2, CMV, EBV and influenza peptides | At Day 0, at the third injection visit and at one month after the last injection
Structure and specificity of the TCR (T-cells Receptors) repertoire of blood cells | At Day 0, at the third injection visit and at one month after the last injection
  High throughput TCR sequencing (Barennes et al, Nat Biotech, 2021) will be performed on separated CD8 and CD4 T cells. Standard diversity metrics, such as V and J gene usage, VJ combination and clonotype frequencies will describe the global repertoire structures before and after vaccination. TCR signatures that could characterize the immune response to vaccination will be define based on the dynamics of sequences. For such studies, analyses are based exclusively on the CDR3 region of the TCRs such as to analyze humans independently of their HLA genotype. Finally, we will search for virus specific TCRs using our curated database (Barennes et al, Nat Biotech, 2021)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Pitié-Salpêtrière - AP-HP, Paris, France

REFERENCES:
- [Derived] Louapre C, Belin L, Marot S, Hippolyte A, Januel E, Ibrahim M, Jeantin L, Zafilaza K, Malet I, Charbonnier-Beaupel F, Rosenzwajg M, Soulie C, Marcelin AG, Pourcher V. Three to four mRNA COVID-19 vaccines in multiple sclerosis patients on immunosuppressive drugs: Seroconversion and variant neutralization. Eur J Neurol. 2023 Sep;30(9):2781-2792. doi: 10.1111/ene.15925. Epub 2023 Jun 25. PMID 37310391